CLINICAL TRIAL: NCT07099638
Title: Randomized Factorial Trial of Varenicline With Nicotine Lozenges and a Smartphone Medication Adherence Intervention to Promote Smoking Cessation
Brief Title: Trial of Varenicline With Nicotine Lozenges and a Smartphone Medication Adherence Intervention for Smoking Cessation
Acronym: COMBOII
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Brown University (Other); Thomas Jefferson University (Other); Sidney Kimmel Cancer Center at Thomas Jefferson University (Other); OU Health Stephenson Cancer Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRB Number 17722; R01CA298165 (NIH)
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Varenicline; Nicotine Lozenges; Medication Adherence; Smartphone Intervention
MeSH Terms: conditions — Smoking Cessation; Medication Adherence | interventions — Varenicline; Tobacco Use Cessation Devices; Nicotine Replacement Therapy

STUDY DESIGN:
Intervention Model Description: The study will employ a 2x2 factorial design in which participants will be randomized to combinations of two treatment factors: 1) pharmacological treatment (varenicline + nicotine lozenges vs. varenicline alone) and 2) smartphone medication adherence intervention (smartphone-based smoking cessation app with vs. without adherence components). The primary study outcome will be biochemically confirmed 7-day point prevalence abstinence at 26 weeks after the scheduled quit date.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Varenicline + Smartphone Intervention with adherence components (VAR + ADHERE) (Experimental): Participants will receive 13 weeks of varenicline (1 titration week + 12 weeks at full twice daily 1 mg dosing) and a smartphone-based smoking cessation intervention with medication adherence components. All participants will receive up to 6 telephone counseling calls.
  Interventions: Drug: Varenicline (VAR); Behavioral: Smartphone intervention with adherence components (ADHERE); Behavioral: Telephone Counseling
- Varenicline + Lozenges + Smartphone Intervention with adherence components (VAR + NRT + ADHERE) (Experimental): Participants will receive 13 weeks of varenicline (1 titration week + 12 weeks at full twice daily 1 mg dosing), 12 weeks of nicotine lozenges (2 mg or 4 mg), and a smartphone-based smoking cessation intervention with medication adherence components. All participants will receive up to 6 telephone counseling calls.
  Interventions: Drug: Varenicline (VAR); Drug: Nicotine lozenge (NRT); Behavioral: Smartphone intervention with adherence components (ADHERE); Behavioral: Telephone Counseling
- Varenicline + Smartphone Intervention without adherence (VAR + NO ADHERE) (Experimental): Participants will receive 13 weeks of varenicline (1 titration week + 12 weeks at full twice daily 1 mg dosing) and a smartphone-based smoking cessation intervention without medication adherence components. All participants will receive up to 6 telephone counseling calls.
  Interventions: Drug: Varenicline (VAR); Behavioral: Smartphone intervention without adherence components (NO ADHERE); Behavioral: Telephone Counseling
- Varenicline + Lozenges + Smartphone Intervention without adherence (VAR + NRT + NO ADHERE) (Experimental): Participants will receive 13 weeks of varenicline (1 titration week + 12 weeks at full twice daily 1 mg dosing), 12 weeks of nicotine lozenges (2 mg or 4 mg), and a smartphone-based smoking cessation intervention without medication adherence components. All participants will receive up to 6 telephone counseling calls.
  Interventions: Drug: Varenicline (VAR); Drug: Nicotine lozenge (NRT); Behavioral: Smartphone intervention without adherence components (NO ADHERE); Behavioral: Telephone Counseling

INTERVENTIONS:
Drug: Varenicline (VAR) — 13 weeks of varenicline
Drug: Nicotine lozenge (NRT) — 12 weeks of nicotine lozenges
  Arms: Varenicline + Lozenges + Smartphone Intervention with adherence components (VAR + NRT + ADHERE); Varenicline + Lozenges + Smartphone Intervention without adherence (VAR + NRT + NO ADHERE)
Behavioral: Smartphone intervention with adherence components (ADHERE) — Smartphone-based smoking cessation intervention with adherence components
  Arms: Varenicline + Lozenges + Smartphone Intervention with adherence components (VAR + NRT + ADHERE); Varenicline + Smartphone Intervention with adherence components (VAR + ADHERE)
Behavioral: Smartphone intervention without adherence components (NO ADHERE) — Smartphone-based smoking cessation intervention without adherence components
  Arms: Varenicline + Lozenges + Smartphone Intervention without adherence (VAR + NRT + NO ADHERE); Varenicline + Smartphone Intervention without adherence (VAR + NO ADHERE)
Behavioral: Telephone Counseling — Up to 6 telephone counseling sessions with a tobacco treatment specialist

SUMMARY:
Although the prevalence of smoking has declined among U.S. adults, smoking remains the leading preventable cause of cancer incidence and mortality. Quitting smoking increases life expectancy, and quitting at an earlier age is associated with more years of life gained. Effective pharmacotherapies to aid cessation are available, and the combination of behavioral support with pharmacotherapy optimizes cessation outcomes. Varenicline is an effective, first-line smoking cessation treatment, and recent research has investigated combination pharmacotherapy to improve the modest quit rates observed with monotherapy. The findings of two meta-analyses have indicated that varenicline combined with the nicotine patch was more effective than varenicline alone for smoking cessation However, no published studies to date have evaluated the combined impact of varenicline and oral nicotine replacement therapy (NRT) on smoking cessation in a randomized trial. Oral NRT, such as nicotine lozenges, can provide acute relief from cravings/withdrawal, and offers individuals the flexibility to deliver nicotine quickly, in contrast with the continuous, passive, and slow-acting delivery of the nicotine patch. Nevertheless, in clinical trials of other combination pharmacotherapies, participants' adherence to of oral NRT has been suboptimal, making it difficult to determine whether there is an added benefit. Given the near-ubiquity of smartphone ownership (85% of U.S. adults), it is plausible that smartphone-based medication adherence interventions could have a positive influence on pharmacotherapy adherence and smoking cessation. This investigative team has demonstrated the feasibility and potential efficacy of using combination varenicline plus oral NRT treatment to promote smoking cessation in a pilot factorial randomized trial. Likewise, pilot findings showed that medication adherence and smoking cessation rates were higher among those who received smartphone-based medication reminders than those who did not. The proposed study will enroll 496 adults who smoke cigarettes daily. The study will employ a 2x2 factorial design in which participants will be randomized to one of four combinations of two treatment factors: 1) pharmacological treatment (varenicline + nicotine lozenges vs. varenicline alone) and 2) smartphone medication adherence intervention (smartphone-based smoking cessation app with vs. without adherence components). The primary study outcomes will be biochemically-confirmed 7-day point prevalence abstinence at 26 weeks after a scheduled quit date, and medication adherence over the 13-week treatment period. Smartphone-based daily diaries will be employed to assess daily smoking and medication adherence. Notably, the proposed study will employ entirely remote assessment and treatment delivery strategies. Exploratory analyses will evaluate the potential interaction between medication type and the smartphone adherence intervention, and compare the influences of pharmacological treatment type and the medication adherence intervention on weekly physical symptoms (e.g., withdrawal, medication side effects). The overarching goal of the proposed research is to improve smoking cessation treatment and decrease cancer risk.

DETAILED DESCRIPTION:
Study Overview. The study will employ an efficient 2x2 factorial design in which participants are randomized to one of four combinations of two treatment factors: 1) pharmacological treatment (VAR+NRT or VAR) and 2) smartphone-based smoking cessation intervention with or without medication adherence intervention (ADHERE or NO ADHERE). All participants will receive 13 weeks of varenicline including the standard 1-week pre-quit titration period, with half of participants additionally receiving 12 weeks of nicotine lozenges. Those assigned to the ADHERE group will receive a smartphone intervention app that includes medication adherence components: education, medication reminders, medication tracking, and messages following a missed medication dose. Participants assigned to NO ADHERE will receive a smartphone smoking cessation intervention app that does not include medication adherence components. Participants will be provided with smartphones if they do not have one. All participants, regardless of treatment group assignment will receive telephone counseling with a Tobacco Treatment Specialist from the TTRP. The primary study outcomes will be carbon monoxide (CO)-confirmed 7-day point prevalence abstinence at 26 weeks after the scheduled quit date , and medication adherence during the 12-week treatment period (self-reported weekly). Daily smoking and medication adherence will also be assessed via smartphone.

Randomization Plan. Stratified block randomization, with a small block size, will be used to ensure balance between study arms over time. Randomization will be stratified by sex (male vs. female), race/ethnicity (White vs. minoritized race/ethnicity), and cigarettes smoked per day (<10 vs. ≥10). Participants will be randomized following full study enrollment.

Blinding. Participant blinding is not feasible since participants will be aware of whether or not they are provided with nicotine lozenges (in addition to the varenicline provided to all participants), and they will know whether their smartphone app has medication adherence components.

Intervention Components. Counseling. All participants will be scheduled to receive 6 weekly telephone counseling sessions lasting 15-30 minutes each with an experienced tobacco treatment specialist (TTS) though the TTRP. Counseling sessions will begin one week prior to the scheduled quit date and continue weekly through 4 weeks after the quit date. Consistent with Guideline recommendations, counseling will focus on education, skill-building, and support; and will employ cognitive-behavioral and motivational strategies. Topics include benefits of quitting, mood/stress management strategies, making positive lifestyle changes, coping skills, and planning for future challenges. Several recommended strategies will be employed to maintain and evaluate treatment fidelity (e.g., counseling checklists, session duration, and total sessions completed). Participant perceptions of nonspecific counselor characteristics will be assessed. Differences between groups on counseling factors may be included in analyses as covariates.

Varenicline. All participants will be evaluated by a study physician via telephone or video conferencing for eligibility to use varenicline. If appropriate, varenicline will be prescribed and filled through a campus Pharmacy and mailed to participants. During the week prior to the scheduled quit date, participants will begin taking varenicline. Doses will be titrated during the first week of medication use (days 1-3: 0.5 mg once daily; days 4-7: 0.5 mg twice daily) and will continue at 1 mg twice daily for 12 additional weeks. Participants will be advised to continue taking varenicline, even if they return to smoking.

Nicotine Lozenges. Participants randomized to VAR+NRT will be provided with 5 boxes of nicotine lozenges (108 pieces per box; 540 pieces total) by mail. This quantity provides a supply that supports flexible ad lib dosing, while also supporting optimal dosing based on package recommendations. Participants may request additional lozenges during the first 12 weeks after the scheduled quit date, and additional supply requests will be documented. Flexible standard nicotine dosing instructions (printed on the package) will be followed. In summary, participants who smoke their first cigarette of the day >30 minutes after waking will be provided with 2 mg lozenges, and those who smoke within 30 minutes of waking will be provided with 4 mg lozenges. Participants will be encouraged to use a lozenge every 1-2 hours during the first 6 weeks after the scheduled quit date, every 2-4 hours during weeks 7-9, and every 4-8 hours during weeks 10-12. Participants will be advised to use ≥9 lozenges per day during the first 6 weeks after the quit date to maximize the likelihood of cessation.

Smartphone App. The study smartphone app will be configured via the Insight Mobile Health Platform. All participants will download the smartphone app, but only those assigned to ADHERE will have access to the medication adherence components. The main menu screen contains treatment topic options and contact information. ADHERE participants will receive scheduled medication reminder prompts each day. All participants will be prompted to complete daily/weekly study assessments (brief daily diaries; weekly, longer, traditional questionnaires).

Mobile Health Platform. The mHealth Technology Shared Resource at the NCI-designated Stephenson Cancer Center developed the Insight mobile health platform which empowers researchers to build, test, and launch technology-based assessment and intervention tools. Applications are developed using state-of-the-art cross-platform design tools.

Intervention Hardware. Hardware will be shipped to participants' home addresses. Participants will be asked to use their own smartphones; however, they will be provided with a smartphone and cellular service if they do not own one, or their phone does not meet the minimum criteria to support the app. Participants who use their own phones will be compensated $20 per month (for 6 months) to defray the costs of phone service. All participants will be provided with a Bedfont iCOquit Smokerlyzer portable Bluetooth breath CO monitor for remote verification of abstinence via smartphone.

Education. All participants will have access to educational topic via the main menu of the app.

Medication Reminders-Varenicline. All participants randomized to the ADHERE intervention (VAR+ADHERE; VAR+NRT+ADHERE) will receive smartphone medication reminders that correspond with the varenicline dosing schedule. Morning (AM) reminders will appear 30 minutes after participants' self-reported typical wake time. Evening (PM) reminders will appear 4.5 hours before bedtime. Follow-up prompts will appear 30 and 60 minutes after the initial reminder if the participant has not yet taken the dose. Following the 3rd and final follow-up prompt, participants will again be asked whether they have take their varenicline (pill). If the participant responds that they have not taken their pill, they will be asked about the main reason they have not taken their pill. Participants will then receive an adherence promotion message that corresponds with their reason for not taking their medication dose.

Medication Reminders-Nicotine Lozenges. Participants randomized to VAR+NRT+ADHERE will receive smartphone-based medication reminders that correspond with standard NRT dosing schedules in addition to varenicline reminders.

After each reminder message, participants will be asked when they last used a nicotine lozenge. Participants who report that they have not used a lozenge in more than 8 hours will be asked about the main reason that they have not used a lozenge. Participants will then receive an adherence promotion message that corresponds with their reason for not using lozenges.

Other App Features. All participants (regardless of treatment group assignment) may also contact study staff directly by telephone. They may access study contact information (email, phone numbers) through the app main menu. This feature allows participants convenient access to study staff when they have questions or concerns about their medications or other aspects of the study. For ADHERE participants, graphical tracking of medication adherence based on daily diary self-reports of varenicline and NRT use will be available, along with descriptive summary information.

Measures. Treatment variables will be assessed via smartphone-based daily diaries to capture the dynamics of daily medication adherence and smoking, withdrawal symptoms, and medication side effects.

Assessment Schedule. All participants will complete app-based assessments on their smartphones. At baseline, participants will complete a longer initial assessment, with weekly follow-up assessments through 12 weeks after the scheduled quit date, and a final follow-up assessment at 26 weeks after the quit date. In addition, participants will be asked to complete brief daily dairy assessments each morning (30 minutes after waking) to assess smoking and other tobacco and cannabis use during the previous day as well as medication adherence and other relevant variables. Participants will be compensated $1 per day for the completion of daily diary assessments over the first 13 weeks of the study (up to up $92). Participants will earn $50 for the completion of the baseline assessment, and an additional $10 per week over the first 13 weeks for completing weekly questionnaires and a CO breath sample submission (up to $130). Participants will earn $50 for the completion of the final follow-up assessment. Participants may earn up to $322 total via reloadable study credit card.

Smoking Abstinence. Self-reported previous day smoking will be assessed daily from 1- week pre-quit through 12 weeks post-quit, and past 7-day smoking status will be self-reported weekly and at the final follow-up reflecting a commonly used self-report measure of abstinence. Breath sample submissions for biochemical verification of abstinence will be prompted as part of each weekly smartphone assessment and the final follow-up assessment. Participants will submit breath samples via the iCOquit breath CO monitor that connects with their study smartphone via Bluetooth. Participants will be considered abstinent if they report complete abstinence from smoking during the past 7 days and provide a CO breath sample of ≤6 ppm consistent with abstinence. The primary outcome measure is biochemically verified, 7-day point prevalence smoking abstinence at 26 weeks post-quit-date (i.e., 3 months after the end of treatment) per current recommendations. E-cigarette and other tobacco product use will be assessed and considered in alternate outcomes focused on broader tobacco use abstinence, but the primary outcome will be combustible cigarette abstinence.

Treatment Adherence. An adapted version of the the Adherence to Refills and Medications Scale (ARMS) will be used to assess overall participant adherence to each smoking cessation medication during the previous week. Participants will complete one version that assesses varenicline adherence, and the subset of participants assigned to the NRT groups will also complete an NRT version of the MAQ. The MAQ will be administered weekly through 12 weeks after the scheduled quit date. In addition, participants will complete daily EMAs of their NRT and varenicline use/adherence during the previous day (i.e., daily number of lozenges used, daily varenicline adherence [0, 1, or 2 doses taken]). Finally, completed counseling sessions will be summed.

Other Measures. Measures of sociodemographic characteristics, tobacco use characteristics, health, mental health, substance use, and several hypothesized treatment mediators and moderators will be included. In addition, participants will be asked weekly to choose from a list of physical symptoms (e.g., medication side effects, withdrawal symptoms) that they have experienced during the previous week. Participants will be asked to rate the severity of any symptoms they are experiencing.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide documentation of identity (to prevent fraudulent enrollment) and Oklahoma residence (due to limitations on prescribing to out-of-state residents)
* Reports daily smoking ≥5 cigarettes per day
* Provides a breath CO sample ≥6ppm to verify current smoking
* Willing to schedule a smoking cessation attempt within the next 1-2 weeks
* Willing to abstain from smoking cannabis or other combustible products during the study
* Willing to use varenicline and nicotine lozenges
* Willing to participate in the study for ≈6 months
* Able to demonstrate >6th grade literacy which is necessary to read intervention materials and complete study assessments

Exclusion Criteria:

* History of seizures (varenicline contraindication)
* History of allergic reaction to varenicline
* Pregnant, planning to become pregnant, or currently breastfeeding
* Unwilling or unable to use varenicline or nicotine lozenges for other reasons (e.g., severe dry mouth, past history of severe medication side effects)
* Other medical reasons at the discretion of the prescribing physician (e.g., uncontrolled hypertension, recent myocardial infarction)
* Weekly or more frequent use of combustible cannabis during the past 30 days with a score ≥2 on the Cannabis Use Disorder Identification Test-Short Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 496 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Smoking Abstinence (26 weeks post-quit) | 26 weeks after the scheduled quit day
  Self-reported smoking abstinence over the past 7 days with breath CO≤6 ppm

SECONDARY OUTCOMES:
Medication Adherence (weekly) | Weekly starting on the quit day (for varenicline) or 1-week post-quit (for lozenges) through 12 weeks post-quit.
  Adapted version of the Adherence to Refills and Medications Scale (ARMS). Separate scales will be administered to assess past-week varenicline and nicotine lozenge adherence. The measure assesses participants' ability to correctly administer medication. Scores may range from 8-32, with lower scores indicating better adherence.
Medication Adherence (daily) | Assessments begin 1 week before the quit day (varenicline) or on the quit day (lozenges) through 12 weeks post-quit.
  Smartphone daily diary assessments of previous day varenicline and lozenge adherence.
Smoking Abstinence (12 weeks post-quit) | 12 weeks after the scheduled quit day
  Self-reported smoking abstinence over the past 7 days with breath CO≤6 ppm

CONTACTS AND LOCATIONS:
Overall Officials: Darla E. Kendzor, Ph.D., Principal Investigator — The University of Oklahoma Health Sciences; Jasjit S. Ahluwalia, MD, Principal Investigator — Brown University
Locations (1):
- TSET Health Promotion Research Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes